CLINICAL TRIAL: NCT02279901
Title: Impact of Interactive Web-Based Education and Interactive Voice Response (Automated Follow-up) Programs on CPAP Adherence for the Treatment of Obstructive Sleep Apnea
Brief Title: Impact of Automated Education and Follow-up Mechanisms on Patient Engagement
Acronym: EmmiUSleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: ResMed (Industry)
Responsible Party: Principal Investigator, Dennis Hwang, MD, MD, Kaiser Permanente
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: KaiserPermanente; ASMF #104-SR-13 (Other Grant/Funding Number: American Sleep Medicine Foundation)
Record Dates: First submitted 2014-10-28; First posted 2014-10-31 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; CPAP; Continuous positive airway pressure; CPAP compliance; Telemedicine; Automated response mechanisms; Patient engagement; OSA
MeSH Terms: conditions — Sleep Apnea, Obstructive; Patient Participation

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Traditional (No Intervention): Patients will attend a 1 hour OSA Class where OSA education is provided and home sleep testing is set up. These patients return the next day for individual appointments where study is scored and test results are discussed with patient. If study is consistent with OSA based on AHI4% at least 5/hour, patients undergo a 1 week autoCPAP trial. During this week, wireless remote monitoring is performed and troubleshooting is provided via telephone if problems with CPAP use are identified. The autoCPAP is returned during an individual visit, and CPAP is ordered for long-term use based on trial results and patient feedback. Patients are scheduled a 3 month follow-up appointment but are also instructed to call their sleep center case manager prior to that visit if there are problems with CPAP use.
- Telemedicine Education Pathway (Experimental): Patients follow our usual workflow as outlined in the Traditional Pathway. In addition, patients are emailed a link to view the Emmi OSA program within 2 weeks prior to their initial OSA class. If the patient tests positive for OSA and agrees to an autoCPAP trial, the patient is emailed a link to view the Emmi CPAP program. These patients are also scheduled for a 3 month follow-up visit to check CPAP usage.
  Interventions: Behavioral: Telemedicine Education
- Telemedicine IVR Pathway (Experimental): Patients follow our usual workflow as outlined in the Traditional Pathway. Additionally, if CPAP is ordered for long-term therapy, the patient is enrolled into an IVR protocol that automatically analyzes the patient's CPAP use. If specific provider-defined thresholds are met, the platform will automatically deliver feedback messages to the patient (phone call, text messaging, or email) with the intention of encouraging better CPAP use. Patients are instructed to contact the sleep center for any issues with their therapy. This platform also includes a method for patients to track their own usage online. Automated messaging mechanism will be active for 3 months after CPAP is ordered, after which the messaging will stop. These patients are also scheduled for a 3 month follow-up visit.
  Interventions: Behavioral: IVR
- Telemedicine Both Pathway (Experimental): Patients follow our usual workflow as outlined in the Traditional Pathway. In addition, patients are provided both Emmi education programs and IVR follow-up as previously outlined. These patients are also scheduled for a 3 month follow-up.
  Interventions: Behavioral: Telemedicine Education; Behavioral: IVR

INTERVENTIONS:
Behavioral: Telemedicine Education — Emmi Solutions produces Web-based, simple to understand, healthcare related educational programs. These programs are interactive sessions that last about 15 minutes, educating patients on the risk of OSA and assisting in preparing patients for procedures. Two such programs will be sent to patients at preset intervals over the duration of the study:
  1. OSA program
  2. CPAP program
  Links to each of these programs are emailed to the patient and date of birth needs to be verified before the program will start. The programs ask the patient for feedback at regular intervals and provide opportunities throughout to make notes or write down questions that can be later printed. These programs are already approved for clinical use within Kaiser Permanente which has a contract with the vendor.
  Other Names: Emmi
  Arms: Telemedicine Both Pathway; Telemedicine Education Pathway
Behavioral: IVR — Interactive Voice Response (IVR) is a protocol in which automated messages are delivered via e-mail, text or phone to patients to provide feedback regarding their CPAP use, intended to improve therapy adherence. The basic protocol involves the use of CPAP devices that wirelessly send usage data to a cloud platform. Automated algorithms will assess the usage data and send messages to the patient when there is suboptimal usage or excessive leak, or to provide encouragement for successful use.
  Specifically, we will use CPAP devices with built-in modems which will send usage data via cellular network to cloud-based platforms that will automatically analyze the usage data and send the automated messages. Patients also can track their own therapy information through the platform.
  Other Names: U-Sleep; Interactive Voice Response
  Arms: Telemedicine Both Pathway; Telemedicine IVR Pathway

SUMMARY:
The primary and well-known challenge with continuous positive airway pressure (CPAP) is the incomplete adherence of patients to this therapy. Successfully improving CPAP use is likely through emphasizing patient education regarding the risks associated with obstructive sleep apnea (OSA), potential benefits of therapy, teaching techniques to acclimate to CPAP, and providing a system of accountability through a follow-up process. With the changing landscape of healthcare reimbursement which emphasizes achieving positive clinical outcomes, discovering more automated and self-directed methods of educating and follow-up is needed.

The investigators plan to investigate the impact of adjunct Web education and automated follow-up on CPAP use and other measurements of patient engagement. The specific aims of this pilot study are as follows:

1. Assess impact of Telemedicine mechanisms on CPAP use 3 months after initiating therapy in comparison to usual standard of care.
2. Assess impact of Telemedicine mechanisms on functional outcomes and parameters of healthcare utilization at 3 months after initiation of therapy in comparison to usual standard of care.

DETAILED DESCRIPTION:
Background

Obstructive sleep apnea (OSA) is a prevalent condition which based on polysomnographic criteria affects 24% of men and 9% of women in the middle-aged population. Due to its high prevalence, its association with cardiovascular disease, and impact on neurocognitive function such as daytime vigilance, it carries a high healthcare burden in a given population. A recent assessment estimated that the yearly economic cost of OSA to Australia (population around 23 million) to be $21 billion. Thus, it is important for us to consider effective treatment not just for the individual, but cost effective management of the population.

Continuous positive airway pressure (CPAP) therapy remains the gold standard treatment given its ability to provide near-complete physiologic effectiveness regardless of OSA phenotype. This therapy improves daytime vigilance and is currently the only therapy with substantial evidence suggesting improvement in cardiovascular risk. The primary and well-known challenge with CPAP is the incomplete adherence of patients to this therapy (long-term CPAP compliance defined by percentage of days with at least 4 hours usage is typically reported to be around 50%.) Advances in CPAP technology (such as with autoCPAP) have not been shown to enhance use. Rather successfully improving CPAP use is likely through emphasizing patient education regarding the risks associated with OSA, potential benefits of therapy, teaching techniques to acclimate to CPAP, and providing a system of accountability through a follow-up process.

The impact of providing a system of accountability with further education/troubleshooting was reflected in a study showing improved CPAP adherence when usage was tracked daily (through a remote wireless process) followed by a telephone encounter if a problem with CPAP use was revealed. Compared to a control group (usual clinical follow-up), average CPAP use per night was higher (321 minutes versus 207 minutes; p<0.0001) 3 months after initiation of therapy.

The challenge with replicating this telemedicine workflow in a real-world setting is the labor-intensive nature of tracking patients on a daily basis and logistics of dispensing and retrieving wireless modems. Furthermore, patient education is very time-consuming, and the ability to provide comprehensive education without built-in efficiencies could potentially affect the financial health of the provider. With the changing landscape of healthcare reimbursement which emphasizes achieving positive clinical outcomes, discovering more automated and self-directed methods of educating and follow-up is needed.

Web-Based Education

Emmi Solutions produces Web-based, simple to understand, healthcare related educational programs. These programs are interactive sessions that last about 15 minutes, educating patients on the risk of certain medical conditions or assists in preparing patients for procedures. Emmi has also produced OSA related programs:

1. OSA program - this program educates patients on symptoms of OSA, provides animated videos depicting airway narrowing during OSA events, discusses health related risks of OSA such as cardiovascular disease and impact on daytime vigilance, preliminarily discusses CPAP as potential therapy, and discusses the testing process with ambulatory or in-lab polysomnography
2. CPAP program - this program educates patients on how to properly use CPAP and wear the mask, discusses potential benefits of CPAP use including impact on health risks and daytime vigilance, provides methods of acclimating to CPAP, encourages patients to give a dedicated trial of CPAP even if initially having trouble, and instructs on how to care for their device and need to replace equipment.

Links to each of these programs are emailed to the patient and date of birth needs to be verified before the program will start. The programs ask the patient for feedback at regular intervals and provide opportunities throughout to make notes or write down questions that can be later printed. These programs are already approved for clinical use within Kaiser Permanente which has a contract with the vendor.

Interactive Voice Response Interactive Voice Response (IVR) is a protocol in which automated messages are delivered to patients to provide feedback regarding their CPAP use, intended to improve therapy adherence. While IVR refers to voice calls via telephone, we use this term to also include messages that are delivered by text messaging and email. The basic protocol involves the use of CPAP devices that wirelessly send usage data to a cloud platform. Automated algorithms will assess the usage data and send messages to the patient when there is suboptimal usage or excessive leak, or to provide encouragement for successful use (See Figure 1 for programmed thresholds that will trigger a message).

Specifically, the investigators will use CPAP devices with built-in modems (AirSense 10; ResMed Corporation) which will send usage data via cellular network (Verizon or Sprint depending on signal availability) to cloud based platform (AirView; ResMed Corporation). This data will be transferred to a second cloud-based platform (U-Sleep; Umbian), and it is this second platform that will automatically analyze the usage data and send the automated messages back to the patients. With each message, there will be a reminder to contact the sleep center for questions or problems regarding CPAP usage. Patients also have the ability to login to the U-Sleep platform at any time to track their own therapy information.

Study Proposal

The investigators plan to investigate the impact of adjunct Web education and automated follow-up on CPAP use and other measurements of patient engagement. The Kaiser Permanente Fontana Sleep Disorders Center (Fontana, California) is an integrated sleep center that functions as a closed-loop system which balances diagnostic testing with a wide array of different follow-up programs. The primary diagnostic pathway within our center for suspected OSA is with home sleep testing that begins with classroom education and includes setup of home sleep testing device. Subsequent clinical visits are individual appointments, and patients undergo a 1 week autoCPAP trial if OSA is present. If appropriate, patients are subsequently ordered a CPAP for long-term use, and a 3 month follow-up visit is scheduled.

Our study enrolls patients into one of four pathways: 1) One-fourth of our patients will follow our usual workflow that functions as our primary control group (Traditional Pathway); 2) One-fourth will follow the usual workflow with the addition of Emmi OSA education prior to the initial OSA class and Emmi CPAP education in those undergoing an autoCPAP trial (Telemedicine Education Pathway); 3) One-fourth will follow usual workflow with the addition of IVR follow-up (Telemedicine IVR Pathway); 4) One fourth will follow usual workflow with addition of both Emmi programs and IVR follow-up (Telemedicine Both Pathway)

The specific aims of this pilot study are as follows:

1. Assess impact of Telemedicine mechanisms on CPAP use 3 months after initiating therapy in comparison to Traditional pathway patients.
2. Assess impact of Telemedicine mechanisms on functional outcomes and parameters of healthcare utilization at 3 months after initiation of therapy in comparison to Traditional pathway patients.

Methods

Study Design This performance improvement initiative is structured as a randomized controlled trial designed to assess impact of automated educational and follow-up mechanisms on measure of patient engagement in patients with OSA. Consecutive patients triaged to home sleep testing for suspected OSA are scheduled to attend an OSA class (the investigators schedule 5 classes of 13 patients per week). Classes will be variably assigned to follow one of the 4 Pathways (1 Traditional and 3 Telemedicine) thus result in pseudo-randomization effect (classes rather than individual patients are randomized) - See Figure 2. The investigators plan to analyze outcomes between the four pathways after 1000 consecutive patients (anticipated about 250 in each pathway) have attended OSA class and completed their 3 month CPAP follow-up.

Traditional Pathway Patients will attend a 1 hour OSA Class (class size 13) where OSA education is provided and home sleep testing (Nox T3, Carefusion) is set up. These patients return the next day for individual appointments where study is scored and test results are discussed with patient. If study is consistent with OSA based on Apnea Hypopnea Index (AHI4%) at least 5/hour, patients undergo a 1 week autoCPAP trial. During this week, wireless remote monitoring (AirView; ResMed) is performed and troubleshooting is provided via telephone encounter if problems with CPAP use are identified. The autoCPAP is returned during an individual visit, and CPAP is ordered for long-term use based on trial results and patient feedback. Patients are scheduled a 3 month follow-up appointment but are also instructed to call their sleep center case manager (or visit the walk-in clinic) prior to that visit if there are problems with CPAP use.

Telemedicine Education Pathway Patients follow our usual workflow as outlined in the Traditional Pathway. In addition, patients are emailed a link to view the Emmi OSA program within 2 weeks prior to their initial OSA class. If the patient tests positive for OSA and agrees to an autoCPAP trial, the patient is emailed a link to view the Emmi CPAP program. These patients are also scheduled for a 3 month follow-up visit to check CPAP usage.

Telemedicine IVR Pathway Patients follow our usual workflow as outlined in the Traditional Pathway. Additionally, if CPAP is ordered for long-term therapy, the patient is enrolled into an IVR protocol (U-Sleep) that automatically analyzes the patient's CPAP use. If specific provider-defined thresholds are met (Figure 1), the platform will automatically deliver feedback messages to the patient (via patient's choice of phone call, text messaging, or email) with the intention of encouraging better CPAP use. Patients are instructed to contact the sleep center for any issues with their therapy. This platform also includes a method for patients to track their own usage online. Automated messaging mechanism will be active for 3 months after CPAP is ordered, after which the messaging will stop. These patients are also scheduled for a 3 month follow-up visit.

Telemedicine Both Pathway Patients follow our usual workflow as outlined in the Traditional Pathway. In addition, patients are provided both Emmi education programs and IVR follow-up as previously outlined. These patients are also scheduled for a 3 month follow-up.

Measured Variables Age, gender, body mass index, polysomnography respiratory parameters, ESS (Epworth Sleepiness Scale), Functional Outcomes of Sleep Questionnaire - 10 Questions (FOSQ-10) will be assessed at baseline. CPAP use, Epworth sleepiness Scale, and FOSQ-10 will be assessed at 3 month follow-up. These measured variables are already part of our standard clinical assessment. The investigators will also evaluate measures of patient engagement and cost-effectiveness of care by collecting information regarding adherence and number of provider encounters.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of obstructive sleep apnea (OSA)
* Appropriate for home sleep testing
* No prior use of CPAP or other therapies for OSA

Exclusion Criteria:

* Commercial drivers
* Complex sleep disorders (e.g. CSA)
* No DME (durable medical equipment) insurance coverage
* Declines CPAP therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1873 (Actual)
Dates: Start 2014-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Average hours of CPAP use per night: experimental pathway vs. traditional pathway | 3 months
  Difference in 3 month CPAP use (hours per night) between each telemedicine (experimental) pathway compared to the traditional (control) pathway

SECONDARY OUTCOMES:
Average hours of CPAP use per night: experimental pathway vs. experimental pathway | 3 months
  Difference in 3 month CPAP use (hours per night) between each telemedicine pathway (experimental) as compared to other telemedicine (experimental) pathways
ESS (Epworth Sleepiness Score) | 3 months
  Difference in 3 month change in ESS among pathways
FOSQ-10 (Functional Outcomes of Sleep Questionnaire - 10 Questions) | 3 months
  Difference in 3 month change in FOSQ-10 among pathways
Adherence to provider encounters | 3 months
  Difference in encounter no-show rates and percentage of moderate-severe OSA patients that agree to long-term CPAP therapy among pathways
Healthcare utilization | 3 months
  Difference in measures of healthcare utilization (e.g. number of provider encounters, primary care visits, number of patient pharmaceutical prescription fills) among pathways

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Hwang, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- Sleep Center; Fontana Medical Center, Kaiser Permanente, Fontana, California, United States

IPD SHARING:
Plan to Share IPD: No
This study has been conducted solely within Kaiser Permanente, and it is unnecessary to release IPD to external sources or organizations.

REFERENCES:
- [Background] Young T, Palta M, Dempsey J, Skatrud J, Weber S, Badr S. The occurrence of sleep-disordered breathing among middle-aged adults. N Engl J Med. 1993 Apr 29;328(17):1230-5. doi: 10.1056/NEJM199304293281704. PMID 8464434
- [Background] The Economic Cost of Sleep Disorders in Australia. Sleep Health Foundation. Deloitte Access Economics. 2010.
- [Background] Fox N, Hirsch-Allen AJ, Goodfellow E, Wenner J, Fleetham J, Ryan CF, Kwiatkowska M, Ayas NT. The impact of a telemedicine monitoring system on positive airway pressure adherence in patients with obstructive sleep apnea: a randomized controlled trial. Sleep. 2012 Apr 1;35(4):477-81. doi: 10.5665/sleep.1728. PMID 22467985
- [Background] Hwang, Dennis. Pathway to Progress: Kaiser Permanente rethinks its sleep center delivery care model. Sleep Review Magazine. October 2012.
- [Derived] Hwang D, Chang JW, Benjafield AV, Crocker ME, Kelly C, Becker KA, Kim JB, Woodrum RR, Liang J, Derose SF. Effect of Telemedicine Education and Telemonitoring on Continuous Positive Airway Pressure Adherence. The Tele-OSA Randomized Trial. Am J Respir Crit Care Med. 2018 Jan 1;197(1):117-126. doi: 10.1164/rccm.201703-0582OC. PMID 28858567